CLINICAL TRIAL: NCT00302692
Title: "Effects of Beta-Blockade on Cardiovascular Morbidity and Mortality in Elderly Trauma Patients: A Prospective Randomized Clinical Trial"
Brief Title: Use of Beta Blockers in Elderly Trauma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHA 0465044Y
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Multiple Trauma; Cardiovascular Diseases; Aged
MeSH Terms: conditions — Multiple Trauma; Cardiovascular Diseases | interventions — esmolol; Metoprolol

INTERVENTIONS:
Drug: Esmolol
Drug: Metoprolol

SUMMARY:
Advances in medical care have increased the proportion of elderly Americans and enabled them to remain more physically active. This has resulted in an unprecedented increase in the number of geriatric patients admitted to trauma centers. The elderly constitute 23% of trauma center admissions, but 36% of all trauma deaths. This disproportionately high mortality is attributable to a higher prevalence of pre-existing conditions, particularly, cardiac disease. Multi-system injuries result in critical cardiac stress. Although beta-blockade has been shown to decrease morbidity and mortality in patients at risk for myocardial infarction after elective surgery, their use in trauma patients with potential underlying cardiac disease has not been previously studied. We hypothesize that routine administration of beta-blockers after resuscitation will reduce morbidity and mortality in elderly trauma patients with, or at risk for, underlying cardiac disease.

This study is a randomized, prospective clinical trial. One cohort will receive routine trauma intensive care, and the other, the same care plus beta-blockade after completion of resuscitation. The primary outcome will be mortality. Secondary outcomes include MI, length of stay, organ dysfunction, cardiac, and other complications.

Changes in outcome may not be due to reduction in myocardial oxygen demand and heart rate. Laboratory studies demonstrate that circulating inflammatory cytokines contribute to cardiac risk in trauma patients, and their production is influenced by adrenergic stimulation. We will measure circulating IL-6, TNF alpha, IL-1beta, and measure NF-kB and p38 MAP kinase activation in peripheral blood leukocytes, and determine the effect of beta-blockade on the production of these inflammatory markers.

Finally, the wide variation in patient response to beta-blockers is attributed to genetic variability in the adrenergic receptor. Therefore, we will identify single nucleotide polymorphisms (SNPS) within the beta-adrenergic receptor, and determine their effects on mortality and response to beta-blockade. This study will provide the first randomized, prospective trial designed to reduce morbidity and mortality in elderly trauma patients at risk for cardiac disease. The laboratory and genetic component will provide additional insights that may explain treatment effects, lead to new therapeutic strategies, and have the potential to lead to additional areas of investigation.

DETAILED DESCRIPTION:
Methods of Proposed Research

1. Study Design: Prospective, randomized clinical trial.
2. Study Overview: All trauma patients admitted to the ICU > 55 years of age with a primary diagnosis of injury will be screened on admission as study candidates. Patients will be excluded if they have non-survivable injuries, are receiving comfort care only, have an advanced directive limiting aggressive care, heart block, severe asthma, bradycardia (< 60 bpm), are on beta-blocker therapy, or are having an acute or evolving myocardial infarction. Informed consent will be obtained. Some patients may be unable to provide consent. In such cases, consent will be obtained from legal surrogates. Consented patients will be randomized into an experimental or control group. Study procedures will commence when end-points of resuscitation have been met for 12 hours, defined as cessation of transfusion and fluid bolus requirements, a systolic blood pressure > 100 mm Hg, heart rate < 130 bpm, adequate urine output, and a resolving base deficit. The experimental group will receive beta-blockers adjusted to keep heart rate 60-80 bpm from the end of resuscitation to hospital discharge. A formal algorithm has been developed for this purpose, and will be inserted into the admission order sheet. Briefly, this will be achieved initially by titration of intravenous esmolol hydrochloride until the patient remains at goal heart rate on a stable dose for 24 hours, then with IV or PO metoprolol. Therapy will be withheld in the event of hypotension (< 100 mmHg), or decreased cardiac index (< 2.0 L/min/m2) accompanied by signs of inadequate end-organ perfusion. The control group will receive the standard of care for the injured geriatric patient. Such patients are not routinely provided with beta-blocker therapy. However, beta-blockers will be used for treatment of excessive tachycardia, dysrhythmias, and post myocardial infarction management, as clinically indicated.
3. Baseline Data Collection: Will include; age, gender, demographic information, co-morbid conditions, pre-injury medications, mechanism of injury, Injury Severity Score, Abbreviated Injury Severity Score (AIS). In our intensive care unit, pulmonary artery catheters are routinely inserted in critically injured elderly trauma patients who do not respond to initial resuscitation. Patients with a PAC will have a complete hemodynamic profile (PAWP, CVP, MAP, PAM, CI, SV, SVRI, PVRI, LVSWI) and O2 transport profile (SvO2, DO2I, VO2I) recorded. Laboratory studies will include serum lactate, base deficit, CBC, electrolytes, and coagulation profile. Blood will also be obtained to measure baseline levels of markers of inflammation (IL-6, IL-1, TNF), cardiac injury (troponin), as well as for peripheral blood leukocyte isolation for measurements of p38 MAP kinase and NF-kB activation, and genotyping.
4. Resuscitation and Daily Management: Our intensive care unit is a closed unit staffed by a group of six dedicated faculty, all of whom have certification in critical care. Treatments, including resuscitation end-points, management of fluid/electrolytes, ventilator therapy, weaning, evaluation/treatment of fever/sepsis, pain/sedation, nutrition, as well as management of specific injury types, are provided according to established clinical protocols, thus reducing or eliminating treatment bias and potentially confounding management variations.
5. Outcome Measures:

   1. Mortality: The primary outcome will be mortality. All patients will be followed from time of enrollment to study completion. Therefore, duration of follow-up will vary from 1-23 months.
   2. Cardiac Events: ICU records (flow charts, labs, ECG) will be screened daily for evidence of dysrhythmia, ischemia/MI, and hypotension. Diagnosis of MI will be based on clinical symptoms, ECG changes, cardiac biomarkers, and autopsy data, if available. Studies on the detection of myocardial infarction demonstrate that incidence is dependent on the type, frequency, and timing of a diagnostic test, as well as the criteria being used. Our study will base the determination of MI on the consensus document of the Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of MI.47 The timing of diagnostic tests will be based on the AHA guidelines for myocardial infarction surveillance for high and intermediate risk patients after major surgical procedures. Accordingly, an ECG will be obtained at baseline, daily for two days, after any surgical procedure, and at ICU discharge. Biochemical markers will be obtained at baseline, after any surgical procedure, daily for two days, and on day 4 or day of ICU discharge (whichever comes first).26 Classification of cardiac events will be done by individuals blinded to group assignment.
   3. Infection/Organ Dysfunction: ICU records will be screened daily for evidence of infection (fever, altered WBC, pneumonia, abdominal abscess, UTI, line sepsis). Sepsis and MOD will be calculated by individuals blinded to group allocation.
   4. Length of Stay: ICU stay, ventilator days, and hospital stay will be recorded.
6. Laboratory Procedures:

   1. Serum Troponins: Serum cardiac troponin I will be determined by ELISA.
   2. Inflammatory Markers: WBC's will be isolated from whole blood by centrifugation, and nuclear proteins isolated to measure NF-kB nuclear translocation. Nuclear protein extracts will be assayed by ELISA with the TransAM NF-kB p65 activation assay to determine the degree of NF-kB activation following LPS stimulation. The amount of translocated NF-kB will be standardized to total protein content, which will be determined in a standard Bradford assay.48 Activation of p38 MAP kinase will be conducted with the p38 MAP kinase assay kit. Briefly, a monoclonal phoso-specific antibody to p38 MAP kinase (Thr180/Tyr182) is used to selectively immunoprecipitate active p38 MAP kinase from the cell lysates. The resulting immunoprecipitate is incubated with ATF-2 fusion protein in the presence of ATP and kinase buffer. This allows immunoprecipitated active p38 MAP kinase to phosphorylate ATF-2. Phosphorylation of ATF-2 at Thr71 is measured by Western blotting using a phosphor-ATF-2 (Thr71) antibody.

      IL-6 concentrations in plasma will be determined by conventional ELISA, using OptEIATM Sets. Briefly, a plate is coated with a monoclonal antibody that is specific for IL-6. Standards and samples are added to the wells, and any IL-6 present binds to the immobilized antibody. The wells are washed and incubated at room temperature with an avidin-horseradish peroxidase conjugate mixed with a biotinylated anti-human IL-6 antibody. The wells are again washed and a TMB substrate solution is added producing a color change. The microwell absorbances are read at 450 nm. The concentration of IL-6 is directly proportional to the color intensity of the test sample.
   3. Sequencing of Beta-Adrenergic Receptor Genotype: The Ser49Gly and Arg399Gly SNP's of the adrenergic receptor will be amplified by polymerase chain reaction (PCR). Genotypes will be assayed by pyrosequencing and DNA sequence analysis. Genomic DNA will be extracted from whole blood by ammonium acetate-ethanol precipitation and the yield quantified by comparison of staining intensity relative to lanes containing known concentrations of standards.49 Fragments containing each of the SNP's will be individually PCR-amplified from genomic DNA using a thermal profile, reaction conditions, and primer sequences specific for each SNP. All genotypes will be determined by pyrosequence analysis using PSQ 96 SNP Software. Each SNP will be assayed with a specific primer sequence, which will enable the scoring of heterozygotes and alternate homozygotes with equal reliability. Amplification conditions have been established and optimized for more than two dozen loci in our laboratory over the past two years. The addition of new candidate SNPs has become a routine matter. We have utilized these protocols to generate genotype data for more than 20 SNP's in over 600 individuals that have been published five manuscripts over the past several years.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients admitted to the ICU > 55 years of age with a primary diagnosis of injury will be screened on admission as study candidates.

Exclusion Criteria:

* Patients will be excluded if they have non-survivable injuries, are receiving comfort care only, have an advanced directive limiting aggressive care, heart block, severe asthma, bradycardia (< 60 bpm), are on beta-blocker therapy, or are having an acute or evolving myocardial infarction.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2005-12; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Mortality
Cardiovascular Morbidity

SECONDARY OUTCOMES:
Inflammatory Profile

CONTACTS AND LOCATIONS:
Overall Officials: Randall Friese, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Derived] Friese RS, Barber R, McBride D, Bender J, Gentilello LM. Could Beta blockade improve outcome after injury by modulating inflammatory profiles? J Trauma. 2008 Apr;64(4):1061-8. doi: 10.1097/TA.0b013e3181684cf0. PMID 18404076